CLINICAL TRIAL: NCT02047032
Title: Effect of Electroacupuncture Versus PFMT Plus Solifenacin for Moderate and Severe Mixed Urinary Incontinence in Female: a Multicenter, Noninferiority, Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture Versus PFMT Plus Solifenacin for Mixed Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Dean of Acupuncture Department of Guangan'men Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012BAI24B01-MUI
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Urinary Incontinence
Keywords: electroacupuncture; urinary incontinence; PFMT; Solifenacin
MeSH Terms: conditions — Urinary Incontinence | interventions — Acupuncture Therapy; Electroacupuncture; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental): BL33 and BL35 of both sides are used. Every session will last for 30 minuets and will be given every other day. There are 36 sessions for each participant in all (3 session per week, 12 weeks).
  Interventions: Procedure: acupuncture
- Solifenacin plus PFMT (Active Comparator): Both PFMT and solifenacin will be given for 36 weeks. Solifenacin will be taken 5mg once daily, before or after meal. PFMT includes intensive exercises conducted in hospital and home exercises. Intensive exercises will be done once every week for the first 12 weeks and once every four weeks for the 13th to 36th week. Home exercises will be done three times daily for 36 weeks.
  Interventions: Drug: solifenacin; Procedure: PFMT

INTERVENTIONS:
Procedure: acupuncture — For BL33, the needle (75mm) will be inserted at the point upper and outside of BL33. Insert the needle with a 30-45°angle to a depth of 50-60 mm. The needle will be manipulated with an even lifting, thrusting and twisting method and the sense of soreness and distention will radiate to the perineal region or the anus. For BL35, the needle will be inserted upward and outward slightly with an even lifting, thrusting and twisting method. The sense of soreness and distention will radiate to the perineal region or the anus. The electric stimulator will be put on the two pair of points with a spare-dense wave, 10/50 Hz, 0.1-5.0 mA. The current intensity will be increased until the participant can not stand.
  Other Names: electroacupuncture
  Arms: acupuncture
Drug: solifenacin — Solifenacin used in this trial is produced by Astellas Pharma Europe B.V.(Country medicine accurate character No. J20090109 )
  Other Names: competitive cholinergic receptor antagonist
  Arms: Solifenacin plus PFMT
Procedure: PFMT — Intensity of the PFMT exercises will conform to the guideline of National Institute for Health and Clinical Excellence (NICE).
  Other Names: pelvic floor muscle training
  Arms: Solifenacin plus PFMT

SUMMARY:
A noninferiority randomized controlled trial aimed at comparing the effect and safety of electroacupuncture versus the pelvic floor muscle training (PFMT) plus solifenacin for mixed urinary incontinence (MUI).

DETAILED DESCRIPTION:
Participants experiencing mixed urinary incontinence will be recruited from 10 centers. A gynecologist or urologist will make the diagnosis. Central randomization will be performed by the Clinical Evaluation Center of the China Academy of Chinese Medical Sciences in Beijing.

Sample size: Sample size is based on the primary outcome. According to literature, the investigators predict that MUI patient's average 72-h incontinence episode frequency of the week 1-12 will decrease by 60% from the baseline after treatment of PFMT plus solifenacin. The number of the acupuncture group is 57%. For the assessment of noninferiority, 250 participants will be needed for each group allowing for a 15% dropout (α=0.05，β=0.2，δ=15%).

Quality control: A 3-level monitoring system (monitors responsible for one center, monitors responsible for all centers and monitors responsible for the whole trial) will be established to check the performance of the trial in time. Outcome assessment, completion of case report forms and data management will be under strict supervision.

Data management: The Remote Dara Capture (RDC) system will be used for data entering. Both paper and electronic case report form will be reserved. A data verification plan is made.

ELIGIBILITY:
Inclusion Criteria:

* females meet the meet the diagnostic criteria of mixed urinary incontinence
* aged 35-75 years
* moderate and severe urinary incontinence with the urinary incontinence severity index between 3 and 9
* suffering from urinary incontinence at least for 3 months with the 72-h incontinence episode frequency≥2 in the baseline assessment
* voluntarily join the research and sign the informed consent

Exclusion Criteria:

* pure stress urinary incontinence, pure urgency urinary incontinence, overflow incontinence and neurogenic bladder
* medicine use for urinary incontinence or may affect the bladder function, or taking any non-drug therapy (such as electric stimulation, bladder training and pelvic floor muscle training) in the last month
* symptomatic urinary tract infection and non-functional urologic disease
* having ever undergone an operation for urinary incontinence or on the pelvic floor (including hysterectomy)
* pelvic organ prolapse degree ≥2
* residual urinary volume (RUV) >30 mL
* maximum flow rate (Qmax) <20 mL/s;
* be allergic to solifenacin or having contradictions for muscarine antagonist (such as urinary retention, gastric retention, myasthenia gravis, ulcerative colitis and angle closure glaucoma)
* diseases affect function of lower urinary tract, such as uncontrolled diabetes, multiple sclerosis, Alzheimer's disease, Parkinson's disease, spinal injury, cauda equina injury and multiple system atrophy.
* serious cardiovascular, pulmonary, cerebral, liver, kidney, hematopoietic system or psychiatric disease and cognitive impairment
* patients with severe renal dysfunction or moderate hepatic dysfunction who are using strong Cyp3a4 Inhibitor like ketoconazole
* unable or limited to walking, up and down stairs and running
* poor compliance with electroacupuncture, pelvic floor muscle training or drug
* pregnancy, lactation or within the 12 months after birth
* having a cardiac pacemaker, a metal allergy, or a severe needle phobia.
* volunteer of other trials

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, doctor, Study Director — Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hargreaves E, Baker K, Barry G, Harding C, Zhang Y, Kandala NB, Zhang X, Kernohan A, Clarkson CE. Acupuncture for treating overactive bladder in adults. Cochrane Database Syst Rev. 2022 Sep 23;9(9):CD013519. doi: 10.1002/14651858.CD013519.pub2. PMID 36148895
- [Derived] Sun B, Liu Y, Su T, Sun Y, Liu Z. Electroacupuncture for stress-related urinary incontinence in elderly women: data analysis from two randomised controlled studies. BMJ Support Palliat Care. 2022 May;12(e1):e164-e170. doi: 10.1136/bmjspcare-2019-002034. Epub 2020 Jan 9. PMID 31919102
- [Derived] Liu B, Liu Y, Qin Z, Zhou K, Xu H, He L, Li N, Su T, Sun J, Yue Z, Zang Z, Zhang W, Zhao J, Zhou Z, Liu L, Wu D, Wu J, Zhou J, Pang R, Wang Y, Liu J, Yu J, Liu Z. Electroacupuncture Versus Pelvic Floor Muscle Training Plus Solifenacin for Women With Mixed Urinary Incontinence: A Randomized Noninferiority Trial. Mayo Clin Proc. 2019 Jan;94(1):54-65. doi: 10.1016/j.mayocp.2018.07.021. PMID 30611454
- [Derived] Liu B, Wang Y, Xu H, Chen Y, Wu J, Mo Q, Liu Z. Effect of electroacupuncture versus pelvic floor muscle training plus solifenacin for moderate and severe mixed urinary incontinence in women: a study protocol. BMC Complement Altern Med. 2014 Aug 15;14:301. doi: 10.1186/1472-6882-14-301. PMID 25128002

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture | Solifenacin Plus PFMT
Started | 250 | 250
Completed | 245 | 235
Not Completed | 5 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Solifenacin Plus PFMT | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.11) | 53.7 (9.38) | 54.2 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 250 | 500
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change From Baseline in 72-hour Incontinence Episode Frequency (IEF) Over Weeks 1-12
Description: The average 72-h IEF is calculated based on a 72-h bladder diary. All relevant time points used in the calculation in the Time Frame (baseline, weeks 1-12)
Time Frame: baseline, weeks 1-12
Population: 1 patient withdrew consent and did not receive electroacupuncture treatment, 2 refused to participate and did not receive PFMT-solifenacin treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Electroacupuncture: BL33 and BL35 of both sides are used. Every session will last for 30 minuets and will be given every other day. There are 36 sessions for each participant in all (3 session per week, 12 weeks).
  acupuncture: For BL33, the needle (75mm) will be inserted at the point upper and outside of BL33. Insert the needle with a 30-45°angle to a depth of 50-60 mm. The needle will be manipulated with an even lifting, thrusting and twisting method and the sense of soreness and distention will radiate to the perineal region or the anus. For BL35, the needle will be inserted upward and outward slightly with an even lifting, thrusting and twisting method. The sense of soreness and distention will radiate to the perineal region or the anus. The electric stimulator will be put on the two pair of points with a spare-dense wave, 10/50 Hz, 0.1-5.0 mA. The current intensity will be increased until the participant can not stand.
Arm/Group | Solifenacin Plus PFMT | Electroacupuncture
Number analyzed (Participants) | 248 | 249
percent change | -36.49 [-43.87 to -29.11] | -37.83 [-41.96 to 33.70]

2. Secondary Outcome: Percentage of Change From Baseline in Mean 72-hour IEF During Weeks 13-24 and Weeks 25-36
Description: Calculated as the same way as the primary outcome. But this outcome will be assessed at different time point.
Time Frame: baseline, weeks 13-24, week 25-36
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
percent change
  Weeks 13-24 | -58.20 [-63.19 to -53.22] | -56.69 [-61.77 to -51.61]
  Weeks 25-36 | -64.20 [-68.77 to -59.63] | -65.48 [-70.14 to -60.82]

3. Secondary Outcome: Percentage of Participants With ≥50% Decrease in Average 72-h Incontinence Episode Frequency
Description: Count the number of cases with the reduction of average 72-h incontinence episode frequency ≥50% and divide it by the number of participants at baseline.
Time Frame: Weeks 1-12, 13-24, 25-36
Population: For various reasons, participants discontinued study.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
Participants
  Weeks 1-12: number analyzed (Participants) | 248 | 239
  Weeks 1-12 | 109 | 112
  Weeks 13-24: number analyzed (Participants) | 245 | 235
  Weeks 13-24 | 174 | 164
  Weeks 25-36: number analyzed (Participants) | 245 | 235
  Weeks 25-36 | 190 | 188

4. Secondary Outcome: Change of Episodes From Baseline in Average 72-hour Urgencies/Urination/Nocturia Episodes
Description: The average 72-h IEF (urinary incontinence, stress urinary incontinence and urgency urinary incontinence respectively) is calculated based on a 72-h bladder diary. For example, the average 72-h incontinence episodes from the 13th to 36th week equal to the sum of 72-h incontinence episodes of the 16th, 20th, 24th, 28th, 32nd, 36th weeks divided by 6.
Time Frame: Baseline, weeks 1-12, 13-24, 25-36
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
percent change
  Change in the 72-h urgence, Weeks 1-12 | -2.62 [-3.20 to -2.05] | -2.99 [-3.58 to -2.41]
  Change in the 72-h urgence, Weeks 13-24 | -4.75 [-5.32 to -4.19] | -4.77 [-5.35 to -4.19]
  Change in the 72-h urgence, Weeks 25-36 | -5.55 [-6.12 to -4.97] | -5.55 [-6.14 to -4.96]
  Change in the 72-h urination, Weeks 1-12 | -3.23 [-3.93 to -2.53] | -3.62 [-4.33 to -2.91]
  Change in the 72-h urination, Weeks 13-24 | -5.96 [-6.70 to -5.22] | -5.26 [-6.02 to -4.51]
  Change in the 72-h urination, Weeks 25-36 | -7.02 [-7.85 to -6.19] | -6.11 [-6.96 to -5.26]
  Change in the 72-h nocturia, Weeks 1-12 | -0.79 [-1.01 to -0.50] | -0.87 [-1.08 to -0.65]
  Change in the 72-h nocturia, Weeks 13-24 | -1.38 [-1.60 to -1.15] | -1.33 [-1.56 to -1.11]
  Change in the 72-h nocturia, Weeks 25-36 | -1.58 [-1.79 to -1.36] | -1.58 [-1.80 to -1.36]

5. Secondary Outcome: Change From Baseline in the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) Score
Description: The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF (range, 0 [best]-21 [worst] outcomes, and 2.52 as minimal clinically important differences (MCID)) scores.
Time Frame: baseline, weeks 12, 24 and 36
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
units on a scale
  Week 12 | -3.96 [-4.32 to -3.61] | -3.73 [-4.09 to -3.37]
  Week 24 | -6.44 [-6.90 to -5.98] | -5.97 [-6.44 to -5.50]
  Week 36 | -7.06 [-7.51 to -6.60] | -6.80 [-7.26 to -6.34]

6. Secondary Outcome: Weekly Median Number of Urine Pads Used During Weeks 1-12, 13-24, and 25-36
Time Frame: Baseline, weeks 1-12, 13-24, 25-36
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: urine pads
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
urine pads
  Weeks 1-12 | 8.0 [5.0 to 11.0] | 9.0 [5.0 to 12.0]
  Weeks 13-24 | 7.0 [4.0 to 10.0] | 8.0 [5.0 to 12.0]
  Weeks 25-36 | 8.0 [4.0 to 10.0] | 8.0 [5.0 to 12.0]

7. Secondary Outcome: the Amount of Urine Leakage (Grams) Measured by the 1-hour Pad Test at Weeks 4 and 12
Description: The performance of 1-hour pad test according to the International Incontinence Society:
  Participants were instructed to void 2 hours before the pad test. On arrival, they received a pre-weighed pad and were asked to sit and drink 500 ml sodium-free water in 15 minutes. Next, they were instructed to walk for 30 minutes, including going up and down 24 stairs. On returning to the clinic, the participants were instructed to perform several activities, including standing and sitting 10 times, coughing vigorously 10 times, running for 1 minute, picking up a coin from the floor 5 times, and putting their hands under water for 1 minute. After the activities were completed, the pad was reweighed to measure the amount of urinary leakage using a gram sensitive weight scale (Xiangshan, EK3820).
Time Frame: Weeks 4 and 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: amount of leakage (grams)
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
amount of leakage (grams)
  Week 4 | -6.74 [-7.93 to -5.56] | -6.96 [-8.17 to -5.76]
  Week 12 | -12.16 [-13.18 to -11.15] | -11.49 [-12.52 to -10.46]

8. Secondary Outcome: Patient's Treatment Satisfaction Degree
Description: The self-assessing satisfaction degree on a 5-point Likert scale (range, 1 [unsatisfied strongly] to 5 [satisfied strongly]) will be finished by participants to evaluate their satisfaction for the treatment.
Time Frame: Weeks 12, 36
Population: 1 patient withdrew consent and did not receive electroacupuncture treatment. 2 refused to participate and did not receive PFMT-solifenacin treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Solifenacin Plus PFMT | Electroacupuncture
Number analyzed (Participants) | 248 | 249
Participants
  Week 12: number analyzed (Participants) | 234 | 243
  Week 12: Marked satisfaction | 58 | 62
  Week 12: Satisfaction | 84 | 112
  Week 12: No change | 80 | 56
  Week 12: Dissatisfaction | 12 | 12
  Week 12: Marked dissatisfaction | 0 | 1
  Week 36: number analyzed (Participants) | 234 | 244
  Week 36: Marked satisfaction | 77 | 85
  Week 36: Satisfaction | 90 | 101
  Week 36: No change | 58 | 47
  Week 36: Dissatisfaction | 9 | 11
  Week 36: Marked dissatisfaction | 0 | 0

9. Secondary Outcome: Patient Global Impression Improvement
Description: Participants will be asked to finish one item evaluating their present condition.
Time Frame: Weeks 12, 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
Participants
  Week 12: number analyzed (Participants) | 244 | 234
  Week 12: Marked improvement | 69 | 52
  Week 12: Moderate improvement | 85 | 75
  Week 12: Slight improvement | 82 | 96
  Week 12: No change | 8 | 8
  Week 12: Slight worsening | 0 | 3
  Week 12: Moderate worsening | 0 | 0
  Week 12: Marked worening | 0 | 0
  Week 36: number analyzed (Participants) | 245 | 235
  Week 36: Marked improvement | 87 | 74
  Week 36: Moderate improvement | 93 | 92
  Week 36: Slight improvement | 55 | 59
  Week 36: No change | 9 | 9
  Week 36: Slight worsening | 1 | 1
  Week 36: Moderate worsening | 0 | 0
  Week 36: Marked worening | 0 | 0

10. Secondary Outcome: Electroacupuncture Acceptance Assessment
Description: The acceptance of electroacupuncture will be tested within 5 minute with a 5-point scale ('0' means very difficult to accept and '4' means accept easily). Median of scores of the three times will be calculated.
Time Frame: Weeks 2, 6 and 12
Population: 1 patient withdrew consent and did not receive electroacupuncture treatment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Electroacupuncture
Number analyzed (Participants) | 249
units on a scale
  Week 2 | 3.0 [3.0 to 3.0]
  Week 6 | 3.0 [2.0 to 3.0]
  Week 12 | 3.0 [2.0 to 3.0]

11. Secondary Outcome: The Number of Participants Using Urine Pads
Time Frame: Weeks 1-12, 13-24, 25-36
Population: For various reasons, the participants discontinued study.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
Participants
  Weeks 1-12: number analyzed (Participants) | 248 | 240
  Weeks 1-12 | 86 | 105
  Weeks 13-24: number analyzed (Participants) | 244 | 237
  Weeks 13-24 | 68 | 80
  Weeks 25-36: number analyzed (Participants) | 244 | 237
  Weeks 25-36 | 59 | 72

12. Secondary Outcome: Change of Episodes From Baseline in Mean 72-h Incontinence Episodes
Time Frame: Weeks 1-12, 13-24, 25-36
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Number analyzed (Participants) | 249 | 248
episodes
  Weeks 1-12 | -4.56 [-5.13 to -3.98] | -4.37 [-4.95 to -3.79]
  Weeks 13-24 | -7.27 [-7.83 to -6.70] | -6.95 [-7.52 to -6.37]
  Weeks 25-36 | -8.31 [-8.83 to -7.78] | -8.22 [-8.76 to -7.69]

ADVERSE EVENTS:
Arm/Group | Electroacupuncture | Solifenacin Plus PFMT
Serious Adverse Events (participants affected / at risk) | 0/250 | 1/250
Other Adverse Events (participants affected / at risk) | 41/250 | 90/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electroacupuncture (N=250) | Solifenacin Plus PFMT (N=250)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electroacupuncture (N=250) | Solifenacin Plus PFMT (N=250)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 62 (62)
constipation (Gastrointestinal disorders) | 0 (0) | 7 (7)
stomach (Gastrointestinal disorders) | 1 (1) | 6 (6)
diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (5)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
upper respiratory infection (Reproductive system and breast disorders) | 19 (19) | 10 (10)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 2 (2) | 2 (2)
hypogeusia (Nervous system disorders) | 0 (0) | 2 (2)
blurred vision (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
herpes zoster (Nervous system disorders) | 1 (1) | 0 (0)
low back pain (Nervous system disorders) | 0 (0) | 1 (1)
pruritus (Nervous system disorders) | 0 (0) | 1 (1)
urinary tract infection (Nervous system disorders) | 2 (2) | 0 (0)
dysuria (Nervous system disorders) | 0 (0) | 1 (1)
dry eye (Eye disorders) | 0 (0) | 1 (1)
facial edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
subcutaneous hematoma (Injury, poisoning and procedural complications) | 10 (10) | 0 (0)

LIMITATIONS AND CAVEATS:
The noninferiority margin to PFMT-solifenacin in MUI women was hard to define. PFMT were led by trained research assistants instead of professional therapists, which may dilute the effect of the control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes